CLINICAL TRIAL: NCT05681273
Title: A Phase I Study to Evaluate the Drug-Drug Interaction of Chiglitazar With Empagliflozin，Atorvastatin and Valsartan in Healthy Subjects.
Brief Title: Drug-Drug Interaction Study of Chiglitazar in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CGZ110
Record Dates: First submitted 2022-12-27; First posted 2023-01-12 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2022-12

CONDITIONS: T2DM
MeSH Terms: interventions — chiglitazar; empagliflozin; Atorvastatin; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): D1: Oral single dose of Empagliflozin 10 mg; D5~9: Oral multiple doses of Chiglitazar 48 mg; D10: Oral single dose of Empagliflozin 10 mg and Chiglitazar 48 mg.
  Interventions: Drug: Chiglitazar; Drug: Empagliflozin
- Group B (Experimental): D1: Oral single dose of Atorvastatin 20 mg; D5~9: Oral multiple doses of Chiglitazar 48 mg; D10: Oral single dose of Atorvastatin 20 mg and Chiglitazar 48 mg.
  Interventions: Drug: Chiglitazar; Drug: Atorvastatin
- Group C (Experimental): D1: Oral single dose of Valsartan 160 mg; D5~9: Oral multiple doses of Chiglitazar 48 mg; D10: Oral single dose of Valsartan 160 mg and Chiglitazar 48 mg.
  Interventions: Drug: Chiglitazar; Drug: Valsartan

INTERVENTIONS:
Drug: Chiglitazar — Chiglitazar 48mg
Drug: Empagliflozin — Empagliflozin 10mg
  Arms: Group A
Drug: Atorvastatin — Atorvastatin 20mg
  Arms: Group B
Drug: Valsartan — Valsartan 160mg
  Arms: Group C

SUMMARY:
This Phase 1 open label study is being conducted to characterize the pharmacokinetic (PK) and safety profiles of Chiglitazar with Empagliflozin，Atorvastatin and Valsartan in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between the ages of 18 and 45 years, inclusive;
* 19.0≤BMI≤26.0 kg/m2. Weight of male ≥50 kg and Weight of female ≥ 45 kg.

Exclusion Criteria:

* History of clinically significant allergy or atopic allergic disease, or allergy to the study drug;
* Previous surgery may affect drug absorption, distribution, metabolism and excretion; or have suffered from gastrointestinal, liver and kidney diseases that can affect drug absorption or metabolism in the past 6 months;
* History of tuberculosis;
* Frequent infection history in the past year, or serious infections leading to hospitalization within 3 months before administration;
* untreated diarrhea, or diarrhea within 7 days before administration;
* Any drugs, vitamin products or herbal medicine used within 1 month before administration;
* History of drug abuse;
* Participated in clinical trial within 3 months before administration;
* Blood donation or massive blood loss within 3 months before the first administration;
* Pregnant or lactating women;
* Regular drinking history; or took any alcoholic products within 48 hours before administration; or positive alcohol test;
* Regular smoking history within 3 months before administration or cannot quit smoking during the trial;
* GFR<80 mL/min;
* Abnormal results of laboratory examination,vital signs, 12 lead ECG, physical examination and chest X-ray;
* Systolic blood pressure<90 or ≥ 140 mmHg, diastolic blood pressure<60 or ≥ 90 mmHg;
* Other situations that are not suitable for participate the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Cmax | up to 72 hours
  Maximum plasma concentration
AUC0-t and AUC0-inf | up to 72 hours
  Area under of the curve (AUC0-t and AUC0-inf)

CONTACTS AND LOCATIONS:
Overall Officials: Hongrong Xu, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan hospital, Shanghai, China